CLINICAL TRIAL: NCT06832228
Title: Prospective Single-center Study of Pomalidomide Combination with Rituximab and Anti-PD-1 Antibody （PPR） in Third or Later Line Therapy of Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of Pomalidomide Combination with Rituximab and Anti-PD-1 Antibody （PPR） in Third or Later Line Therapy of DLBCL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPR
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-06

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pomalidomide combination with rituximab and Anti-PD-1 Antibody (Experimental): All patients will receive the PPR regimen (a total of 4-6 cycles, 28 days for each cycle):
  * pomalidomide: 4 mg, orally, once daily from Day 1 to Day 21.
  * Rituximab: 375 mg/m², administered on Day 1.
  * PD-1: 200 mg, administered on Days 1. Patients who achieved PR or CR after 6 cycles were treated with maintenance therapy at the investigator's discretion (1-2 years).
  Interventions: Drug: Pomalidomide Combination With Rituximab and Anti-PD-1 Antibody （PPR）

INTERVENTIONS:
Drug: Pomalidomide Combination With Rituximab and Anti-PD-1 Antibody （PPR） — All patients will receive the PPR regimen (a total of 4-6 cycles, 28 days for each cycle):
  * pomalidomide: 4 mg, orally, once daily from Day 1 to Day 21.
  * Rituximab: 375 mg/m², administered on Day 1.
  * PD-1: 200 mg, administered on Days 1.

SUMMARY:
This study aims to observe and explore the efficacy and safety of pomalidomide combination with rituximab and Anti-PD-1 Antibody in Third or Later Line Therapy of diffuse large B-cell lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily joined the study, signed the informed consent, and had good compliance;
* Patients with 18 Years to 80 Years(at the time of signing the informed consent); Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score: 0-2;
* Patients with histopathologically confirmed diffuse large B-cell lymphoma with evaluable lesions who did not achieve CR or relapsed after second-line therapy
* Female patients of reproductive age should agree that birth control (such as intrauterine device, birth control pills, or condoms) must be used during the study period and for six months after completion; Having a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating; Male patients should agree to use contraception during the study period and for six months after the end of the study.

Exclusion Criteria:

* Pathological subtypes: primary central nervous system DLBCL or primary mediastinal large B-cell lymphoma.
* Presence of severe or uncontrolled comorbid conditions including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, active peptic ulcer disease, or severe hemorrhagic disorders such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring transfusion or other medical interventions.
* A history of any active immune or autoimmune disease, or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Any active infection requiring systemic antimicrobial therapy within 14 days before starting study treatment, including, but not limited to, bacterial, fungal, and viral infections.
* Current participation in other clinical studies, or initiation of study drugs administration less than 4 weeks after completion of previous clinical study treatment.
* Patients with concomitant diseases that, in the investigator's judgment, may seriously endanger patients' safety or may interfere with the completion of the study, or are deemed unsuitable for inclusion for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 28days after the end of treatment
  The proportion of subjects who achieves a best overall response of CR or PR.

SECONDARY OUTCOMES:
Complete Remission Rate（CRR） | 28days after the end of treatment
  The proportion of subjects who achieves a best overall response of CR.
Disease-control Rate（DCR） | 28days after the end of treatment
  The proportion of subjects response of CR, PR, or SD
Progression-Free Survival（PFS） | Up to 2 years
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first
overall survival（OS） | Up to 2 years
  The overall survival time refers to the time from therapy to death due to any cause.
Adverse event rate | From date of first day of treatment until 30 day after last treatment
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Yang, PhD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No